CLINICAL TRIAL: NCT03841838
Title: The Effect of Energy Drink on Cardiovascular Variables: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 19-03
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
Keywords: Energy drink; Heart rhythm; QT prolongation; Blood pressure
MeSH Terms: conditions — Cardiovascular Diseases; Long QT Syndrome | interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Energy drink (Experimental): Two 12 oz bottles of energy drink
  Interventions: Other: Energy drink
- Placebo (Placebo Comparator): Two 12 oz bottles of placebo drink
  Interventions: Other: Placebo drink

INTERVENTIONS:
Other: Energy drink — Two 12 oz bottles of commercially available energy drink
  Arms: Energy drink
Other: Placebo drink — Two 12 oz bottles placebo drink. Placebo drink will contain carbonated water, lime juice, and cherry flavoring.
  Arms: Placebo

SUMMARY:
Many adults in the United States regularly consumer energy drinks. Currently, the safety of energy drinks is still questionable and there are many reports associating energy drinks with adverse events including hospitalizations and deaths. Previous research shows that energy drink can affect heart rhythm and elevate blood pressure. However, these studies use a higher volume (32 ounces) of energy drinks than those available in the market (24 ounces). The purpose of this study is to study if 24-ounce energy drinks can significantly affect heart rhythm and elevate blood pressure when compared to a placebo.

DETAILED DESCRIPTION:
The study is a randomized, double blind, controlled, crossover study comparing the effect of energy drinks and placebo on cardiovascular parameters including heart rhythm and blood pressure.

Subjects who contact the PI for interest in study participation will be scheduled a time to study facility for initial evaluation on eligibility criteria. At initial evaluation, participants will be informed about the study details, presented with Informed Consent Document (ICD), and be asked to sign the appropriate forms voluntarily if they decide to participate. Once consented, participants will be asked a series of questions and screened for blood pressure and heart rhythm parameters to determine eligibility to enroll. If patient is eligible to enroll, they will be allocated a randomized identification number.

Participants will be randomly assigned to consume either two-12 oz bottles of energy drink and two-12 oz bottles of control drink on 2 separate days. The study will occur over approximately 8 days with each session taking about 5 hours per day. Each session will have 6 days between each other.

Participants will be expected to refrain from any products containing caffeine or alcohol 48 hours and fast 10 hours before each study visit. At the beginning of each study visit, baseline measurements of ECG, blood pressures, and heart rate will be obtained prior to consuming study drinks. Repeat measurements will be obtained every 60 minutes after consumption over 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults 18-40 years old
* Participants must be willing to refrain from caffeine and alcohol use 48 hours prior to each study day
* Participants must be willing to fast 10 hours prior to each study day
* Participants must have health insurance

Exclusion Criteria:

* Corrected QT (QTc) interval greater than 450 milliseconds (ms). QTc will be determined on the ECG obtained during initial screening appointment.
* Blood pressure at initial screening appointment greater than 140/90 mmHg.
* Presence of any known medical condition confirmed through participant interview
* Concurrent use of ANY medication taken on a daily basis, to include herbal products or supplements (exception include oral contraceptives that will be allowed if taking for longer than 1 month)
* Current smokers or those who have smoked any cigarettes within the past month
* Pregnant or currently breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
QTc interval | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in QTc interval from baseline in each of 2 arm
Central systolic blood pressure | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in central systolic blood pressure from baseline in each of 2 arm

SECONDARY OUTCOMES:
QT interval | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in QT interval from baseline in each of 2 arm
PR interval | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in PR interval from baseline in each of 2 arm
QRS duration | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in QRS duration from baseline in each of 2 arm
Heart rate | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in heart rate from baseline in each of 2 arm
Central diastolic blood pressure | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in central diastolic blood pressure from baseline in each of 2 arm
Peripheral systolic and diastolic blood pressure | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in peripheral systolic and diastolic blood pressures in each of 2 arm
Augmentation index | Measurements are obtained at baseline and every 60 minutes after study drink consumption over 4 hours
  Maximum change in augmentation index from baseline in each of 2 arm

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Lee, PharmD, Principal Investigator — University of the Pacific
Locations (1):
- University of Pacific, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher EA, Lacey CS, Aaron M, Kolasa M, Occiano A, Shah SA. Randomized Controlled Trial of High-Volume Energy Drink Versus Caffeine Consumption on ECG and Hemodynamic Parameters. J Am Heart Assoc. 2017 Apr 26;6(5):e004448. doi: 10.1161/JAHA.116.004448. PMID 28446495
- [Background] Shah SA, Occiano A, Nguyen TA, Chan A, Sky JC, Bhattacharyya M, O'Dell KM, Shek A, Nguyen NN. Electrocardiographic and blood pressure effects of energy drinks and Panax ginseng in healthy volunteers: A randomized clinical trial. Int J Cardiol. 2016 Sep 1;218:318-323. doi: 10.1016/j.ijcard.2016.05.007. Epub 2016 May 13. PMID 27240158
- [Background] Shah SA, Chu BW, Lacey CS, Riddock IC, Lee M, Dargush AE. Impact of Acute Energy Drink Consumption on Blood Pressure Parameters: A Meta-analysis. Ann Pharmacother. 2016 Oct;50(10):808-15. doi: 10.1177/1060028016656433. Epub 2016 Jun 23. PMID 27340146
- [Background] Phan JK, Shah SA. Effect of caffeinated versus noncaffeinated energy drinks on central blood pressures. Pharmacotherapy. 2014 Jun;34(6):555-60. doi: 10.1002/phar.1419. Epub 2014 Mar 19. PMID 24644139
- [Background] Hajsadeghi S, Mohammadpour F, Manteghi MJ, Kordshakeri K, Tokazebani M, Rahmani E, Hassanzadeh M. Effects of energy drinks on blood pressure, heart rate, and electrocardiographic parameters: An experimental study on healthy young adults. Anatol J Cardiol. 2016 Feb;16(2):94-9. doi: 10.5152/akd.2015.5930. Epub 2015 Mar 23. PMID 26467367
- [Background] Elitok A, Oz F, Panc C, Sarikaya R, Sezikli S, Pala Y, Bugan OS, Ates M, Parildar H, Ayaz MB, Atici A, Oflaz H. Acute effects of Red Bull energy drink on ventricular repolarization in healthy young volunteers: a prospective study. Anatol J Cardiol. 2015 Nov;15(11):919-22. doi: 10.5152/akd.2015.5791. Epub 2015 Mar 5. PMID 25868042